CLINICAL TRIAL: NCT04324242
Title: Activating Transversus Abdominis Muscle: A Comparison Of Two Different Feedback Methods
Brief Title: Activating Transversus Abdominis Muscle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Esra Dülger, Research Assistant, Hacettepe University
Other Study IDs: GO 16/808
Record Dates: First submitted 2020-03-24; First posted 2020-03-27 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-04

CONDITIONS: Low Back Pain; Rehabilitative Ultrasound; Spinal Stabilization
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1: visual feedback
  Interventions: Other: abdominal hallowing maneuver
- Group2: traditional feedback
  Interventions: Other: abdominal hallowing maneuver

INTERVENTIONS:
Other: abdominal hallowing maneuver — abdominal hallowing maneuver includes tucking navel in and up. To be able to control the effect of breathing it was instructed to start the maneuver at the end of the expiration. During the maneuver it was instructed to focus on increasing the thickness of TrA without increasing the thickness of IO and EO

SUMMARY:
Transversus abdominis (TrA) is an important muscle for spinal stabilization. Abdominal draw-in maneuver (ADIM) is a method that selectively activates TrA without activating external oblique (EO) and internal oblique (IO) muscles. Individuals with low back pain may have some troubles to understand proper contraction of TrA. Therefore, to contract the TrA, two different feedback techniques have been used to instruct. In this observational study we aim to investigate the effects of two different biofeedback methods to teach patients the proper activation of TrA muscle using ADIM. We aim to find out the differences between visual and traditional tactile biofeedback and decide which one is practical and easy to teach the patients in clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers between ages of 18-25

Exclusion Criteria:

* Volunteers excluded if they had (1) history of LBP, (2) spinal or abdominal surgeries, (3) neuromusculer or romatologic diseases. Each volunteer gave their informed consent.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers between ages of 18-25 with no spinal problems.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-04-13 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-09-15 (Estimated)

PRIMARY OUTCOMES:
thickness change in TrA muscle | 1 month
  thickness change in TrA muscle

SECONDARY OUTCOMES:
thickness change in EO muscle | 1 month
  thickness change in EO muscle
thickness change in IO muscle | 1 month
  thickness change in IO muscle

CONTACTS AND LOCATIONS:
Overall Officials: Sevil Bilgin, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No